CLINICAL TRIAL: NCT00533364
Title: A Phase I/II Study to Assess the Effect of Soluble Beta-1,3/1,6-glucan in Combination With Standard Therapy in Patients With Breast Cancer
Brief Title: Effect of SBG in Patients With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotec Pharmacon ASA (Industry)
Responsible Party: VP Clinical Development, Biotec Pharmacon ASA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBG-2-01
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: SBG (Soluble beta-glucan) — Oral administration, three dose levels, administered day 1-8 in each 3-weeks treatment cycle, 4 treatments cycles.

SUMMARY:
This study is set up to determine whether soluble beta-glucan (SBG) has

* unfavourable side effects
* beneficial treatment effects when given in combination with standard antibody and chemotherapy to patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histologically/cytologically confirmed locally advanced or metastatic breast cancer
2. Primary tumor or metastases are HER2-ICH3+ or FISH+
3. Measurable or non-measurable disease
4. The patients must not have received treatment with the combination trastuzumab and vinorelbine previously
5. Expected lifetime of more than 12 weeks
6. Age ≥ 18 years
7. Performance status ≤ 2 according to World Health Organization (WHO) scale
8. The patient must be able to comply with the protocol
9. Verbal and written informed consent

Exclusion Criteria:

1. Women who are pregnant or breast-feeding. A negative pregnancy test must be provided during the screening period for fertile women. Fertile women must use effective contraceptive methods
2. Clinical symptoms indicating central nervous system involvement
3. Other current or former malignant disease, with the exception of adequately treated and cured carcinoma in situ cervicis uteri and basocellular skin carcinomas
4. Left ventricular ejection fraction (LVEF) < 50% of normal range
5. Reduced bone marrow function defined by leukocyte counts < 3.0 x 109/l and neutrophil counts < 1.5 x 109/l, or thrombocyte counts ≤ 100 x 109/l
6. Reduced liver function defined by bilirubin > 3 x upper normal limit and/or ASAT/ALAT > 3 x upper normal limit and/or alkaline phosphatase > 3 x upper normal limit.
7. Reduced renal function defined by serum creatinine > 2 x upper normal limit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Asess the safety of SBG in combination with standard antibody and chemotherapy treatment | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erik Wist, MD, PhD, Principal Investigator — Ullevaal University Hospital
Locations (2):
- Norway (2):
  - Ålesund Hospital, Ålesund
  - Ullevål University Hospital, Oslo